CLINICAL TRIAL: NCT00547716
Title: The Effect of Omega-3 Fatty Acids (Omacor@) on the Response Rate to Antiviral Therapy in Patients With Chronic Hepatitis C Infection
Brief Title: Use of Omega-3 Fatty Acids (Fish Oil) in Patients With Chronic Hepatitis C Infection
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of study enrollment.
Sponsor: University of Missouri, Kansas City (Other)
Collaborators: Reliant Pharmaceuticals (Industry); Saint Luke's Health System Foundation (Unknown); Truman Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 07-48
Record Dates: First submitted 2007-10-19; First posted 2007-10-23 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2017-01

CONDITIONS: Hepatitis C
Keywords: Hepatitis C; Omega 3 fatty acids; Omacor; Interferon
MeSH Terms: conditions — Hepatitis C | interventions — Fatty Acids, Omega-3; Omacor

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1. (Experimental): Omega-3 Fatty Acids 4 grams/day
  Interventions: Dietary Supplement: Omega-3 Fatty Acids
- 2. (Placebo Comparator): Placebo comparator along with interferon.
  Interventions: Drug: Placebo comparator

INTERVENTIONS:
Dietary Supplement: Omega-3 Fatty Acids — Omega-3 Fatty Acids - 4 grams per day
  Other Names: Omacor@
  Arms: 1.
Drug: Placebo comparator
  Arms: 2.

SUMMARY:
Hepatitis C virus infection is the most common blood-borne infection in the United States and is a leading cause of chronic liver disease affecting 130 million people around the world. It is estimated that 1.6% of the US population may be affected by Hepatitis C infection. The only recommended treatment that has been approved for your condition is the use of interferon and ribavirin. In patients with chronic Hepatitis C, there tends to be an accumulation of fat in the liver. Fatty liver has been associated with failure of treatment.

The accumulation of fat in the liver has been blamed on a particular type of fat called triglycerides. Fish oil, by reducing a type of fat called VLDL, can lower the triglyceride concentration by as much as 50 percent or more. This study seeks to determine if the administration of fish oil along with standard treatment to patients with Hepatitis C will increase the treatment response rates.

DETAILED DESCRIPTION:
Hepatic steatosis may be present in up to 66% of cases of chronic Hepatitis C infection. Previous studies have reported steatosis to be an independent predictor of treatment failure in patients with chronic hepatitis C infection.

The pathogenesis of hepatic steatosis in chronic Hepatitis C infection has not been fully elucidated. Hepatic steatosis is a manifestation of excessive triglyceride accumulation in the liver. Hypertriglyceridemia may benefit from Omega-3 fatty acid (fish oil supplements) which, by reducing VLDL production can lower the serum triglyceride concentration by as much as 50 percent or more.

The treatment of chronic hepatitis C results in an average sustained viral response rate of 54%-63%. We have found response rates of around 50% on treatment of patients. We hypothesize that by giving omega-3 fatty acids along with interferon therapy for patients with Hepatitis C, we may be able to increase the treatment response rates. Thus, the purpose of the study is to look at the effect of omega 3 fatty acids on early and sustained viral response rates in patients with chronic HCV infection.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients > 18 years of age
* Patients with chronic hepatitis C infection
* Patients receiving interferon for treatment of hepatitis C

Exclusion Criteria:

* pregnant or lactating patients
* End stage target organ damage in diabetes mellitus: advanced renal failure (serum creatinine >2.0 mg/dl) with or without dialysis, severe neuropathy, advanced peripheral vascular disease.
* Anticipated life expectancy less than 2 years
* Co-existent etiologies for liver disease
* Alcohol consumption more than 30 g per day in men and more than 20 g per day in women.
* Patients on Omega-3 fatty acid supplementation or those patients who report eating oily fish such as salmon, albacore tuna, sardines, etc. twice a week or more frequently.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-06; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
To assess whether omega-3 fatty acids can improve early and sustained viral responses to treatment with interferon in patients with chronic infection. | To be determined by Hepatits C genotype

SECONDARY OUTCOMES:
To look at the effect of treatment of Hepatitis C on insulin resistance. | While using Omega-3 Fatty Acid capsules

CONTACTS AND LOCATIONS:
Overall Officials: Laura M Alba, M.D., Principal Investigator — Truman Medical Center; Jagdish Nachnani, MD, Principal Investigator — Truman Medical Center
Locations (2):
- United States (2):
  - Truman Medical Center, Kansas City, Missouri
  - Saint Luke's Hospital, Kansas City, Missouri

REFERENCES:
- See also: Hepatitis information — http://www.cdc.gov/Ncidod/diseases/hepatitis/c/index.htm